CLINICAL TRIAL: NCT01657773
Title: Study of the Prevalence of Colorectal Cancer in Patients With Nonalcoholic Fatty Liver Disease.
Brief Title: Study of the Association of Nonalcoholic Fatty Liver Disease With Colorectal Malignant Neoplasm
Acronym: NWC
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Ming-Hua Zheng, Attending physician, Wenzhou Medical University
Other Study IDs: wenzhouMC 001
Record Dates: First submitted 2012-07-29; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Neoplasms; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Colorectal Neoplasms; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- colorectal cancer, without nonalcoholic fatty liver disease: Patients were performed colonoscopy examination for colorectal cancer and who had been foud colorectal cancer proven by biopsy.Then the colorectal cancer patients who had not been diagnosed with nonalcoholic fatty liver disease was based on blood tests and abdomen ultrasound examination.
  Interventions: Other: Ultrasound examination and Colonoscopy examination
- colorectal cancer, with nonalcoholic fatty liver disease: Patients were performed colonoscopy examination for colorectal cancer and who had been foud colorectal cancer proven by biopsy.Then the colorectal cancer patients who had been diagnosed with nonalcoholic fatty liver disease was based on blood tests and abdomen ultrasound examination ultrasonography.
  Interventions: Other: Ultrasound examination and Colonoscopy examination

INTERVENTIONS:
Other: Ultrasound examination and Colonoscopy examination

SUMMARY:
The aim of this sudy is to investigate the prevalence of colorectal cancer (CRC) in patients with nonalcoholic fatty liver disease (NAFLD) and evaluate whether NAFLD is a risk factor for CRC.

DETAILED DESCRIPTION:
As one of the most common cancer worldwide, colorectal cancer (CRC) is a major cause of cancer death in Asian countries. And during the past three decades, the incidence of CRC has been increasing rapidly in china. Many studies supported that cigarette smoking, obesity and insulin resistance were associated with CRC. In recent years, metabolic syndrome (MetS) - Including glucose tolerance, dyslipidemia, obesity, hypertension and chronic inﬂammation - and its individual components have been proven to be the risk for colorectal neoplasm. Colonoscopy is the most accurate technique for diagnosis, surveillance and exclusion of colorectal neoplasm for high-risk CRC groups. Therefore, improved risk stratiﬁcation knowledge of the target population is necessary to improve CRC patients' prognosis.

Nonalcoholic fatty liver disease (NAFLD) is the most prevalent chronic liver disease worldwide and cause a wide spectrum of liver damage, such as steatohepatitis, cirrhosis, even end-stage liver disease and hepatocellular carcinoma. NAFLD has been found to be associated with obesity, insulin resistance, hypertension and dyslipidemia, and is considered as a liver manifestation of MetS. Although it has been also well established that MetS and its individual components are risk factors for colorectal neoplasm, as above, there is paucity of research looking at the relation between NAFLD and CRC. Therefore, the investigators aimed to investigate the prevalence of CRC in patients with NAFLD and evaluate whether NAFLD is an independent risk factor for CRC.

ELIGIBILITY:
Inclusion Criteria:

* Patients had colonoscopy and
* Patients had conventional inspections(blood routine, liver function test and abdomen B ultrasonography)

Exclusion Criteria:

* Patients were excluded with history of colorectal cancers or polyps, other extraintestinal malignancies and contraindications to colonoscopy.
* Patients were excluded who had viral hepatitis, cirrhosis, liver cancer or other liver disease.
* Patients ere excluded who drank more than 20g alcohol per day.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted entirely of outpatients. Patients were offered to perform colonoscopy for CRC screening according to the American College of Gastroenterology recommendations. Based on blood tests and abdomen B ultrasonography, patients without NAFLD were regarded as healthy controls and those with NAFLD constituted the community NAFLD cohort. Patients were included only if they had colonoscopy and conventional inspections (blood routine, liver function test and abdomen B ultrasonography). Among them who with history of colorectal cancers or polyps, other extraintestinal malignancies and contraindications to colonoscopy were excluded. Besides, we excluded patients who had viral hepatitis, cirrhosis, liver cancer or other liver disease.Patients who drank more than 20g alcohol per day were also excluded.
Sampling Method: Probability Sample
Enrollment: 2315 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Ultrasound examination | Up to 10 months
  Hepatic ultrasonography scanning was performed on all patients by experienced radiologists who were blinded to the aims of the study and clinical details of the patients. NAFLD was diagnosed by the following criterion: hepatomegaly, the echogenicity of liver parenchyma increased diffusely, and vascular blurring.
Colonoscopy examination | Up to 10 months
  Before performed colonoscopy examination, all patients were given 4L polyethelyne glycol lavage solution for bowel preparation.
  The colonoscopic features include the types, location, size, number of lesions and differentiation of neoplasm.
Statistical analysis | Up to 07 months
  The Binary logistic regression analysis was applied to assay the correlation between NAFLD and CRC after adjustment for independent factors, including age, gender, smoking, and family history.

SECONDARY OUTCOMES:
Patients' baseline characteristics | Up to 10 months
  Patients' baseline characteristics were collected before colonoscopy examination. Smoking, alcohol consumption, past medical history, and family history were all recorded using a standardized questionnaire.Blood pressure (BP) was measured in rest state with a standard mercury sphygmomanometer.
Laboratory Assay and Measurement | Up to 10 months
  Complete blood count, liver function, blood glucose , blood lipids, Cancer Embryo Antigen (CEA) and other related test were performed when underwent colonoscopy examination. The liver function test included alanine aminotranferase, aspartate aminotranferase, albumin, serum sodium, serum chloride, serum chloride and creatinine. Complete blood count was made up of platelet and hemoglobin (Hb). Blood lipids test contains, total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides. Additionally, CEA was detected by conventional serological assays.

CONTACTS AND LOCATIONS:
Overall Officials: MingHua Zheng, Medical Master, Study Chair — First Affiliated Hospital of Wenzhou Medical College; XianFeng Lin, Medical undergraduate, Principal Investigator — Wenzhou Medical University; KeQing Shi, Medical Master, Principal Investigator — First Affiliated Hospital of Wenzhou Medical College; WenYue Liu, Medical undergraduate, Principal Investigator — First Affiliated Hospital of Wenzhou Medical College
Locations (1):
- Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Lin XF, Shi KQ, You J, Liu WY, Luo YW, Wu FL, Chen YP, Wong DK, Yuen MF, Zheng MH. Increased risk of colorectal malignant neoplasm in patients with nonalcoholic fatty liver disease: a large study. Mol Biol Rep. 2014 May;41(5):2989-97. doi: 10.1007/s11033-014-3157-y. Epub 2014 Jan 22. PMID 24449368